CLINICAL TRIAL: NCT02860624
Title: Efficacy and Safety of Ilaprazole for GERD: A Randomized, Double-Blind, Esomeprazole-Controlled, Phase 3, Multicenter Trial in China
Brief Title: Ilaprazole for the Treatment of Gastroesophageal Reflux Disease (GERD) in Chinese Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Livzon Pharmaceutical Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Livzon-IY-81149R-11-01
Record Dates: First submitted 2016-07-26; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-07

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — ilaprazole; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 10 mg ilaprazole (Experimental)
  Interventions: Drug: 10 mg ilaprazole
- 40 mg esomeprazole (Active Comparator)
  Interventions: Drug: 40mg esomeprazole

INTERVENTIONS:
Drug: 10 mg ilaprazole — Two 5-mg ilaprazole tablets (Livzon Pharm Group Inc., China) being taken orally each morning on an empty stomach for 8 weeks
  Arms: 10 mg ilaprazole
Drug: 40mg esomeprazole — One 20-mg omeprazole capsule (AstraZeneca, Losec) being taken orally each morning on an empty stomach for 8 weeks
  Arms: 40 mg esomeprazole

SUMMARY:
This study is designed to evaluate the efficacy and tolerability of ilaprazole relative to that of esomeprazole in healing erosive esophagitis and resolving accompanying symptoms of GERD.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patients will be eligible for enrollment if they:
* are 18-70 years of age,
* have at least one of the two symptoms, heartburn and reflux,
* have photographically documented erosive esophagitis confirmed by esophagogastroduodenoscopy(EGD), and graded according to the Los Angeles (LA) Classification (A-D), within 5 days before randomization to treatment. Female patients are required to be nonpregnant, nonlactating, postmenopausal, surgically sterilized, or using a medically acceptable form of birth control, as determined by the investigator. Women of child- bearing potential will receive a pregnancy test.

Exclusion Criteria:

* Patients will be ineligible if they:
* have cancerous or peptic ulcers, Zollinger-Ellison syndrome, varices of esophagus or fundus of stomach
* have a known history of gastric acid suppression operation, esophageal operation or peptic operation other than simple closure of perforation,
* have severe complications, severe other diseases of digestive tract such as Crohn's disease and ulcerative colitis, and severe other systemic diseases,
* have taken proton pump inhibitors within the 5 days or for more than three consecutive days within the two weeks immediately preceding start of study drug,
* participated in a clinical trial with an investigational drug or device within the past three months,
* have hypersensitivity or idiosyncratic reaction to ilaprazole, esomeprazole or any other benzimidazole,
* have alcoholic intemperance, drug addiction or any other improper habits.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2011-12; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Changes in stage of the ulcer assessed by endoscopic(week 8) changes relative to baseline (week 0) levels. | week 8

REFERENCES:
- [Derived] Xue Y, Qin X, Zhou L, Lin S, Wang L, Hu H, Xia J. A randomized, double blind, controlled, multi center study of Ilaparazole in the treatment of reflux esophagitis-Phase III clinical trial. Contemp Clin Trials. 2018 May;68:67-71. doi: 10.1016/j.cct.2018.03.004. Epub 2018 Mar 11. PMID 29540336